CLINICAL TRIAL: NCT00752401
Title: VITA-D: Cholecalciferol Substitution in Vitamin D Deficient Kidney Transplant Recipients: A Randomized, Placebo-controlled Study to Evaluate the Posttransplant Outcome
Brief Title: Vitamin D3 Substitution in Vitamin D Deficient Kidney Transplant Recipients
Acronym: VITA-D
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Kyra Borchhardt, Priv.-Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VitaD-1; EudraCT Number 2008-002807-21
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Kidney Transplantation; Vitamin D Deficiency; Renal Osteodystrophy
Keywords: Vitamin D; Cholecalciferol; Vitamin D3; 25-hydroxyvitamin D3; Immunomodulation; Vitamin D deficiency; Kidney transplantation; Renal transplantation; Graft function; Acute rejection; Renal osteodystrophy; Posttransplant bone loss
MeSH Terms: conditions — Vitamin D Deficiency; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 6800 IU/day of Cholecalciferol (Vitamin D3) orally for one year
  Interventions: Drug: Cholecalciferol
- 2 (Placebo Comparator): Oral placebo solution daily for one year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — 6800 IU of Cholecalciferol will be administered in the form of Oleovit® D3-drops once a day for one year. Treatment starts on day 5 after kidney transplantation. At serum calcium levels >2,65 mmol/l vitamin D3 administration will be reduced to 3600 IU per day. If calcium levels persist above 2,85 mmol/l over a period of four weeks vitamin D3 administration will be discontinued and restarted when serum calcium levels declined to ≤ 2,65 mmol/l with only 3600 International Units per day.
  Other Names: Vitamin D3; Oleovit® D3
  Arms: 1
Drug: Placebo — An oral placebo solution matching Cholecalciferol in terms of appearance, smell and taste will be administered once a day for one year. Treatment starts on day 5 after kidney transplantation.
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the effects of Cholecalciferol (Vitamin D3) substitution on the posttransplant outcome (glomerular filtration rate as well as serum creatinine levels, number of acute rejection episodes, number of infections and C-reactive protein levels within the first year after transplantation) in vitamin D deficient kidney transplant recipients.

DETAILED DESCRIPTION:
Apart from its classical actions in calcium homeostasis, vitamin D acts as a potent immunomodulatory agent. As such, vitamin D is thought to have beneficial effects in the transplant setting, especially in kidney transplant recipients considering the fact that approximately 40% of all kidney transplant recipients are vitamin D deficient.

Therefore, the objective is to conduct a randomized, double-blind, placebo-controlled study focusing on the impact of Cholecalciferol substitution in vitamin D deficient kidney transplant recipients on graft function (glomerular filtration rate as well as serum creatinine levels), incidence of acute rejection episodes, frequency and severity (CRP levels) of posttransplant infections within the first year after kidney transplantation.

Moreover, the impact of Vitamin D3 on renal osteodystrophy will be analyzed by means of bone mineral density. DXA measurements will be performed during the first four weeks after kidney transplantation, after 5, and after 12 months posttransplant.

Kidney transplant recipients found to have vitamin D deficiency (defined as 25-hydroxyvitamin D < 50 nmol/l) will be included and will be randomized to receive either oral Vitamin D3 therapy or placebo. Vitamin D3 will be administered at a daily dose of 6800IU over a time period of one year.

All in all, 200 subjects will be included in the VITA-D study.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* deceased donor kidney transplant recipients
* only kidney transplant recipients
* vitamin D deficiency defined as 25 (OH)D < 50nmol/l

Exclusion Criteria:

* re-transplantation for the second time if the patient is highly immunized and therefore included in the aphaeresis program
* re-transplantation for the third or further time
* significant impaired intestinal resorption: malabsorption due to celiac sprue, systemic scleroderma; maldigestion due to chronic pancreatitis, pancreatic insufficiency, pancreas resection, mucoviscidosis, Zollinger-Ellison-syndrome
* history of inflammatory bowel disease: Crohn's disease, ulcerative colitis
* previous gastrectomy, small bowel or large bowel resection, intestinal bypass surgery
* severe liver disease: cirrhosis
* HIV positive

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-05; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
The immunologic effects of Vitamin D3 substitution in vitamin D deficient kidney transplant recipients will be evaluated by means of: Glomerular filtration rate | one year after kidney transplantation
Number of acute rejection episodes | one year after kidney transplantation
Number of infections | one year after kidney transplantation
CRP levels | one year after kidney transplantation
Courses of calcium levels | within the first year after kidney transplantation

SECONDARY OUTCOMES:
The impact of Vitamin D3 substitution on renal osteopathy will be analyzed by means of absolute bone mineral density (g/cm2) | within the first year after kidney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Kyra Borchhardt, MD, Principal Investigator — Medical University of Vienna, Department of Internal Medicine III, Division of Nephrology and Dialysis
Locations (1):
- Medical University of Vienna, Department of Internal Medicine III, Division of Nephrology and Dialysis, Vienna, Austria

REFERENCES:
- [Derived] Thiem U, Heinze G, Segel R, Perkmann T, Kainberger F, Muhlbacher F, Horl W, Borchhardt K. VITA-D: cholecalciferol substitution in vitamin D deficient kidney transplant recipients: a randomized, placebo-controlled study to evaluate the post-transplant outcome. Trials. 2009 May 29;10:36. doi: 10.1186/1745-6215-10-36. PMID 19480654